CLINICAL TRIAL: NCT05625438
Title: Bedside Telerehabilitation Early After Stroke
Brief Title: Telerehabilitation Early After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TRCare, Inc. (Industry)
Collaborators: Providence St. Jude Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRC-08
Record Dates: First submitted 2022-11-01; First posted 2022-11-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bedside Telerehabilitation (Experimental): Participants will be assigned 45-minute therapy training exercises each day for 5 days per week.
  Participants will use the HandyMotion device to interact with the telerehabilitation program displayed on the TV set in the patient room.
  Interventions: Device: HandyMotion Treatment Program

INTERVENTIONS:
Device: HandyMotion Treatment Program — A pair of sensor-based wireless remote controllers to allow the performance of functional exercises and games that target arm movement.

SUMMARY:
The goal of this clinical trial is to assess the safety and feasibility of providing extra doses of rehabilitation therapy for persons with a recent stroke. The therapy treatment targets to improve arm function by introducing telerehabilitation to the bedside of participants during the inpatient rehab admission period. Participants will use a newly developed functional training system (HandyMotion) to access therapy treatment program directly from their hospital room. HandyMotion is a sensor-based training system that can connect to the TV set in the hospital room, enabling patients to access their therapy training program to practice rehab-oriented games and exercises ad libitum, at any time of the day.

DETAILED DESCRIPTION:
This clinical trial is designed to address 3 specific aims:

Aim 1: To measure the safety of daily bedside telerehabilitation.

Aim 2: To measure the feasibility of daily bedside telerehabilitation.

Aim 3: To derive a preliminary estimate of motor and functional outcomes in patients engaged in daily bedside telerehabilitation.

Telerehabilitation therapy is delivered over the course of the inpatient rehabilitation stay. A therapist-facing web portal is used for treatment planning and patient monitoring. The treatment approach was initially designed based on an upper-extremity task-specific training manual and Accelerated Skill Acquisition Program.

Each daily 45-minute treatment session is created by a licensed OT or PT and includes:

A. At least 15 min/day of upper extremity exercises. In addition, therapists have the option to incorporate standard exercise equipment (e.g., Theraband or dowels) that can be incorporated into assigned exercises.

B. At least 15 min/day of functional training through games. The study provides 2 controllers with 5 different input devices that are available to drive game play. Games stress various motor control features (e.g., varying movement speed, range of motion, target size, extent of visuomotor tracking, or level of cognitive demand), which are selected and adjusted by the therapist.

C. Five minutes/day of stroke education. The education content targets five categories (Stroke Risk Factors, Stroke Prevention, Effects of Stroke, Diet, and Exercise) and corresponds to the Stroke Knowledge Exam.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Stroke that is radiologically verified, due to ischemia or to intracerebral hemorrhage, and with time of stroke onset <30 days prior to enrollment; or traumatic brain injury.
3. Unilateral arm motor deficits that are neither trivial (no arm weakness) or devastating (arm plegia). This requires that the baseline Box & Block Test score with affected arm to be at least 1 block in 60 seconds but no more than 90% of the number of blocks with the good arm.
4. Possess enough arm movement to participate in therapy
5. Informed consent signed by the subject
6. Able to follow simple instructions
7. Study participation is not likely to be significantly limited by agitated behavior

Exclusion Criteria:

1. A major, active, coexistent neurological or psychiatric disease that would limit study participation, e.g., advanced dementia
2. Expectation that patient's cognitive status will likely interfere substantially with playing assigned games or exercises
3. Deficits in communication that interfere with reasonable study participation
4. Lacking visual acuity, with or without corrective lens, of 20/50 or better in at least one eye
5. Subject does not speak sufficient English to comply with study procedures
6. Shoulder pain that in the judgement of the study team is likely to substantially limit the amount of telerehabilitation therapy completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety of daily beside telerehabilitation based on incidence of treatment-emergent adverse events as assessed by regular review of the medical record and patient interview | "For approximately 2 weeks, up until 2 days prior to discharge"
  Safety will be measured in terms of adverse events (AEs) deemed related to use of the telerehabilitation system on a probable or definite basis.

SECONDARY OUTCOMES:
Feasibility of daily bedside telerehabilitation based on measurement of patient compliance, as determined by reviewing electronic records of device usage | "baseline" and "immediately after end of treatment"
  Feasibility will be measured in terms of patient compliance, specifically the fraction of days where a patient is assigned to do bedside telerehabilitation and initiates a treatment session. Any factors related to reduced compliance, including technical and medical factors, will be recorded.
Box and Blocks Test | "baseline" and "immediately after end of treatment"
  Measure of Upper Extremity Function by assessing unilateral gross manual dexterity. Participant will be asked to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Covarrubias-Eckardt, MD, Principal Investigator — Providence St. Jude Medical Center
Locations (1):
- Providence St. Jude Medical Center, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No